CLINICAL TRIAL: NCT07015268
Title: Phase III Confirmatory Study of KLH-2109 in Patients With Endometriosis
Brief Title: A Clinical Study of KLH-2109 in Patients With Endometriosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KLH1301; Under registration (Other: jRCT)
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — linzagolix; Leuprolide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KLH-2109 group (Experimental): Oral administration
  Interventions: Drug: KLH-2109
- Leuprorelin group (Active Comparator): Subcutaneous administration
  Interventions: Drug: Leuprorelin acetate

INTERVENTIONS:
Drug: KLH-2109 — - KLH-2109 tablet: Oral administration
  - Leuprorelin acetate placebo: Subcutaneous administration
  Arms: KLH-2109 group
Drug: Leuprorelin acetate — - KLH-2109 placebo tablet: Oral administration
  - Leuprorelin acetate: Subcutaneous administration
  Arms: Leuprorelin group

SUMMARY:
To verify the non-inferiority of KLH-2109 to leuprorelin acetate in a double-blind manner in terms of efficacy in endometriosis patients with pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

Premenopausal women aged 18 years or older (at the time of consent) with endometriosis who meet any of the following inclusion criteria.:

* A diagnosis of endometriosis by laparotomy or laparoscopy within 5 years before the start of the screening period;
* Ovarian chocolate cyst confirmed by MRI performed within 1 year before the start of the screening period or ultrasonography (transvaginal, transabdominal, or transrectal) carried out at the start of the screening period; or
* Any of induration of the pouch of Douglas, limitation of uterine mobility, and pelvic tenderness based on the result of pelvic/rectal examination at the start of the screening period and a diagnosis of clinical endometriosis

Exclusion Criteria:

1. Patients with undiagnosed abnormal genital bleeding
2. Patients with abnormal uterine bleeding or anovulatory bleeding judged to be severe by the principal investigator or subinvestigator
3. Patients with concomitant chronic abdominal pain not attributable to endometriosis (such as irritable bowel syndrome [IBS] and interstitial cystitis)
4. Patients with concomitant pelvic inflammatory disease or a history of pelvic inflammatory disease within 8 weeks before obtaining informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the maximum NRS score for pelvic pain during 28 days prior to 12 weeks of the investigational product treatment | 12 weeks
  NRS score for pelvic pain:
  The NRS score for pelvic pain is an integer scale of 0 to 10 in which the worst daily pain associated with endometriosis is scored as 0 for "no pain" and 10 for "the worst pain imaginable."

SECONDARY OUTCOMES:
Change from baseline in and actual values of the maximum NRS score for pelvic pain every 28 days | Up to 24 weeks
  The NRS score for pelvic pain is an integer scale of 0 to 10 in which the worst daily pain associated with endometriosis will be scored as 0 for "no pain" and 10 for "the worst pain imaginable."
Change from baseline in and actual values of the maximum severity score for pelvic pain every 28 days | Up to 24 weeks
  The severity of pelvic pain will be assessed on a five-point scale, based on the most severe pain experienced during the day: as score 0 for "None: No pain", score 1 for "Very mild: Not bothersome, score 2 "Mild: Concerned but tolerable (not requiring analgesics), score 3 for "Moderate: Unbearable (requiring analgesics), and score 4 for "Severe: Intolerable despite the use of analgesics.
Change from baseline in and actual values of severity score for temporary pain at each evaluation time point | Up to 24 weeks
  Pain in bowel movement will be assessed on a five-point scale: as score 0 for "None: No pain", score 1 for "Very mild: Not bothersome", score 2 "Mild: Concerned but tolerable", score 3 for "Moderate: Unbearable to continuously receive stimulation causing the pain", and score 4 for "Severe: Intolerable unless stimulation causing the pain is immediately discontinued".
  Pain during a pelvic examination will be assessed on a four-point scale: as score 0 for "None: No findings", score 1 for "Mild: Pelvic tenderness", score 2 for "Moderate: Between Mild and Severe", and score 3 for "Severe: Severe pelvic tenderness".
  Dyspareunia will be assessed on a five-point scale: as score 0 for "None: No pain", score 1 for "Very mild: Not bothersome", score 2 for "Mild: Feeling pain but tolerable", score 3 for "Moderate: Severe pain and discontinuation due to pain", and score 4 for "Severe: Unbearable severe pain and avoidance of sexual intercourse from the beginning".
Change from baseline in and actual values of severity score of objective findings at each evaluation time point | Up to 24 weeks
  * The severity of the induration of the pouch of Douglas will be assessed on a four-point scale: as score 0 for "None: No findings", score 1 for "Mild: Presence of a small finger-sized induration", score 2 for "Moderate: Between Mild and Severe", and score 3 for "Complete occlusion of the pouch of Douglas with no elasticity".
  * The severity of the limitation of uterine mobility will be assessed on a four-point scale: as score 0 for "None: No findings", score 1 for "Mild: Limited mobility ", score 2 for "Moderate: Severely limited mobility", and score 3 for "Severely limited mobility, no movement at all".
Percent change from baseline in and actual values of ovarian chocolate cyst volume at each evaluation time point | Up to 24 weeks
  The presence or absence of ovarian chocolate cyst in both ovaries will be determined by ultrasonography (transvaginal, transabdominal, or transrectal) and the long and short axes of all ovarian chocolate cysts (unit, mm) will be measured.
Change from baseline in and actual values of EHP-30 domain score at each evaluation time point | Up to 24 weeks
  The EHP-30 is a questionnaire rating scale of 30 items related to QOL in patients with endometriosis on a 5-point scale: "Never", "rarely", "sometimes", "often" and "always". The subjects themselves will evaluate their QOL for the prior month using the EHP-30 questionnaire form and record the results of their assessment in the questionnaire form.
Incidence of adverse events and treatment-related adverse events | Up to 24 weeks
Percent change from baseline in bone mineral density at each evaluation time point | Up to 24 weeks
Change from baseline in T-score at each evaluation time point | Up to 24 weeks
  The "T-score" is an important indicator used in bone density tests. It shows how much an individual's bone density deviates from the average value of young adults (YAM: Young Adult Mean) in terms of standard deviations (SD). Specifically, it is evaluated as follows:
  * -1.0 or above: Normal
  * Between -1.0 and -2.5: Low bone mass (osteopenia)
  * -2.5 or below: Osteoporosis

CONTACTS AND LOCATIONS:
Overall Officials: Yoshitaka Shimizu, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Research Site, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: Yes
* The Individual Patient Data (IPD) are available upon reasonable request and with permission of Kissei Pharmaceutical Co., Ltd.
  * For a data sharing request for IPD, please contact Kissei Pharmaceutical at rinsyousiken@pharm.kissei.co.jp.
Supporting Information: Study Protocol, SAP